CLINICAL TRIAL: NCT00906243
Title: Phase I/IIa Study of RNActive®-Derived Therapeutic Vaccine in Advanced or Metastatic Hormone Refractory Prostate Cancer
Brief Title: RNActive®-Derived Therapeutic Vaccine
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study Closed after completion of Phase I
Sponsor: University of Florida (Other)
Collaborators: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-9103-002
Record Dates: First submitted 2009-05-14; First posted 2009-05-21 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-02

CONDITIONS: Hormone Refractory Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CV9103 (Experimental): CV9103 will be applied intradermally on three (3) or five (5) time points. Treatment with CV9103 is administered over a period of either seven (7) or twenty-three (23) weeks.
  Interventions: Biological: CV9103

INTERVENTIONS:
Biological: CV9103 — CV9103 encodes for 4 prostate specific antigens.

SUMMARY:
This is a Phase I/IIa open, uncontrolled, prospective study, to be conducted in an out-patient setting. The present study is one of two clinical trials of the RNActive®-derived vaccine CV9103 being conducted concurrently in the US and Europe, which represent the first clinical trials conducted for this novel vaccine.

The Phase I part of the study consists of a staggered inclusion of subjects in two cohorts of 3, to confirm the safety of the intended dose (320 µg RNA per antigen), with a lower dose to be considered in case of dose-limiting toxicity (DLT) being reported in greater than or equal to 2 out of 3-6 subjects; in this way, the recommended dose (RD) for the Phase IIa part of the study will be established. In the Phase IIa part of the study, additional subjects will be included at the RD, to confirm the safety and explore the activity of that dose.

DETAILED DESCRIPTION:
Medical Need:

At present, no curative therapy is available for subjects with advanced or metastatic prostate cancer. Approximately 1 of every 3 men present with advanced or metastatic disease; therefore, current standard therapies are ineffective and new therapeutic approaches are warranted. There is ample evidence that active immunotherapy against cancer is safe and capable of stimulating potentially therapeutic immune responses in the cancer patient. Moreover, several Phase II immunotherapy trials have suggested clinical benefit by reducing the tumor mass or prolonging time to progression in subjects with advanced prostate cancer.

Potential Benefits:

CV9103 is an mRNA-based vaccine for the treatment of human prostate cancer that is based on CureVac's RNActive® technology. CV9103 encodes for 4 prostate specific antigens. Because these antigens are present in prostate cancer cells, they are appropriate targets for intervention. These antigens have been shown to correlate frequently with the progression of prostate cancer, and are known to be immunogenic in humans, where they induce antigen specific T-cell or B cell expansion.

As an RNA-based vaccine, CV9103 features several advantages over other approaches: it is highly specific, there is no restriction to the patient's MHC genotype, and it does not need to cross the nuclear membrane to be active. Finally, in the absence of reverse transcriptase, RNA can not be integrated into the genome.

CV9103 will be administered in 5 doses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented history of hormone refractory prostate cancer as evidenced by three consecutive increases in serum PSA despite continued androgen ablative therapy. Serum testosterone levels must be less than 50 ng/dl
* Signed informed consent in accordance with Good Clinical Practice (GCP) and local regulatory requirements prior to trial participation
* Age greater than or equal to 18 yrs (Phase I and IIa) and less than or equal to 75 yrs (Phase IIa only)
* ECOG (Eastern Cooperative Oncology Group) Grade of 0 or 1
* Adequate Hematologic Function with:

  * WBC ≥ 3000 mm3
  * hemoglobin ≥ 10mg/dl
  * platelets ≥ 100,000/mm3
* Adequate Renal and Hepatic Function with:

  * serum creatinine ≤ 1.5 x Upper Limit of Normal
  * bilirubin < 2.0 mg/dl
* Adequate Coagulation Parameters with:

  * Prothrombin INR < 1.5
  * Partial Thromboplastin Time < 1.5 x Institutional Upper Limit of Normal
* Subjects will be advised to use barrier contraception while enrolled in the study and for one month after the last immunization.
* Life Expectancy > 6 month

Exclusion Criteria:

* Subjects who have received radiation therapy within 8 weeks of pretreatment evaluation. (There must be at least 12 weeks if prior therapy included 89-Strontium between any prior therapy and study entry.)
* Subjects who have received chemotherapy, radiation therapy or biologic regimens within 8 weeks of pretreatment evaluation.
* Subjects treated with any investigational agent within the past 30 days are excluded.
* Subjects who have received active immunotherapy, such as Antigen Loaded Dendritic Cells, are excluded (Phase I only). In Phase IIa, Subjects who have received an active immunotherapy based on any of the antigens used in this study either as DNA, RNA or a protein/peptide-based vaccines are excluded. Subjects who have received any other active immunotherapy, such as Antigen Loaded Dendritic Cells, within 6 months prior to study entry are also excluded.
* Subjects who have not recovered from radiation, chemotherapy, or immunotherapy toxicities.
* Subjects with either previously irradiated or new CNS (central nervous system) metastases. (Pre-enrollment head CT is not required.)
* Subjects with a history of autoimmune disease such as, but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis.
* Subjects with serious intercurrent chronic or acute illness such as pulmonary [asthma or chronic obstructive pulmonary disease (COPD)] or cardiac (NYHA class III or IV) or hepatic disease or other illness considered by the P.I. to constitute an unwarranted high risk for investigational drug treatment.
* Medical or psychological impediment to probable compliance with the protocol.
* Concurrent second malignancy other than non-melanoma skin cancer, or controlled superficial bladder cancer. In the event of prior malignancies treated surgically, the subject must be considered NED (no evidence of disease) for a minimum of 3 years prior to enrollment.
* Subjects on steroid therapy (or other immunosuppressive agents such as azathioprine or cyclosporine A) are excluded on the basis of potential immune suppression. Subjects must have had 8 weeks of discontinuation of any steroid therapy prior to enrollment.
* Presence of an active acute or chronic infection, including symptomatic urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot) or viral hepatitis (as determined by HBsAg and Hepatitis C serology).
* Subjects with penicillin allergies

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Vieweg, MD FACS, Principal Investigator — Univeristy of Florida, College of Medicine
Locations (1):
- University of Florida, College of Medicine, Gainesville, Florida, United States

REFERENCES:
- [Derived] Fotin-Mleczek M, Duchardt KM, Lorenz C, Pfeiffer R, Ojkic-Zrna S, Probst J, Kallen KJ. Messenger RNA-based vaccines with dual activity induce balanced TLR-7 dependent adaptive immune responses and provide antitumor activity. J Immunother. 2011 Jan;34(1):1-15. doi: 10.1097/CJI.0b013e3181f7dbe8. PMID 21150709
- See also: Department Website — http://www.urology.ufl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6 subjects entered Phase 1 of the study between June 2009 and December 2009.
Period: Overall Study
Arm/Group | CV9103
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CV9103
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 69.1 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Assessment of Safety and Tolerability of the Trial Regimen
Description: Dose Limiting Toxicity (DLT) is defined as the following treatment-related adverse events or laboratory abnormalities, graded according to NCI-CTCAE version 3.0:
  1. All Categories equal or greater than grade 3
  2. Allergy/autoimmunity equal or greater than grade 2
  3. Dosing delay greater than 48 hours due to toxicity All adverse events will be graded and documented according to Common Terminology Criteria for Adverse Events version 3.0.
Time Frame: At Nine Weeks with Follow Up at One Year
Population: Phase 1 consisted of cohort 1 with 3 subjects and cohort 2 with three subjects.
Measure: Number; unit: events
Arm/Group | CV9103
Number analyzed (Participants) | 6
events | 6

ADVERSE EVENTS:
Arm/Group | CV9103
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CV9103 (N=6)
Erythema (General disorders) | 6 (6) — Injection Site Reaction.
Induration (General disorders) | 6 (6) — Injection Site Reaction
Fatigue (General disorders) | 2 (2) — Administrative Site Condition
Influenza Like Illness (General disorders) | 1 (1) — Administrative Site Conditions
Oedema Peripheral (General disorders) | 1 (1) — Administrative Site Conditions
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthraligia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Peripheral motorneuropathy (Nervous system disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Oral Fungal Infection (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Weight Decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ordpharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruitus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Neopasm Excision (Surgical and medical procedures) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early by decision of the Sponsor after 6 subjects had been enrolled in the Phase I part of the study. No efficacy evaluations were planned during the Phase I part of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This was a Phase 1 and Phase 2 study. The study was terminated after completion of Phase 1 under terms of a settlement agreement that restricts disclosure to limited Phase 1 results only.